CLINICAL TRIAL: NCT05127915
Title: A Prospective, Multicenter, Pivotal Study With Randomized Controlled Prophylactic and Independent Therapeutic Cohorts to Evaluate the Safety and Efficacy of an Absorbable Vena Cava Filter for Pulmonary Embolism Prevention
Brief Title: US Pivotal Clinical Study of the Adient Absorbable Filter for the Prevention of Pulmonary Embolism
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adient Medical (Industry)
Collaborators: Avania (Industry); ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PROT-CI2021
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Pulmonary Embolism
Keywords: Vena Cava Filters; Embolic Protection Devices
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data will be reviewed by the Outcomes Assessor for futility at 25% and 50% enrollment. Subsequently at 75% enrollment, the Outcomes Assessor will conduct an interim assessment for potentially stopping the study with overwhelming efficacy of the filter cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Therapeutic (Experimental): The therapeutic arm will include subjects with diagnosed symptomatic VTE (PE and/or DVT). Each subject will receive an Adient absorbable filter to help prevent a subsequent PE. All study subjects will return to the investigation site for the Follow-up Visits at Week 2 (±3 days), Week 10 (±1 week) and Month 9 (±2 weeks). Subjects will be interviewed and examined at each follow-up visit to perform safety and filter status evaluations.
  Interventions: Device: Adient absorbable filter + best practice VTE prophylaxis
- Prophylactic - Test (Experimental): The Prophylactic - Test arm will include subjects who are at transient high risk for PE and do not have diagnosed symptomatic VTE (PE and/or DVT). If randomized into this prophylactic arm, study subjects will receive an Adient absorbable filter to help prevent PE in addition to being administered current best practice PE prevention, namely sequential compression machines, compression stockings, and anticoagulants when indicated. All study subjects will return to the investigation site for the Follow-up Visits at Week 2 (±3 days), Week 10 (±1 week) and Month 9 (±2 weeks). Subjects will be interviewed and examined at each follow-up visit to perform safety and filter status evaluations.
  Interventions: Device: Adient absorbable filter + best practice VTE prophylaxis
- Prophylactic - Control (Active Comparator): The Prophylactic - Control arm will include subjects who are at transient high risk for PE and do not have diagnosed symptomatic VTE (PE and/or DVT). If randomized into this prophylactic arm, study subjects will receive current best practice PE prevention, namely sequential compression machines, compression stockings, and anticoagulants when indicated. All study subjects will return to the investigation site for the Follow-up Visits at Week 2 (±3 days), Week 10 (±1 week) and Month 9 (±2 weeks). Subjects will be interviewed and examined at each follow-up visit.
  Interventions: Device: best practice VTE prophylaxis

INTERVENTIONS:
Device: Adient absorbable filter + best practice VTE prophylaxis — Adient absorbable filter helps prevent PE during an 8 week protection period then gradually breaks down into carbon dioxide and water within 6 to 8 months. The absorbable filter does not require removal.
  Arms: Prophylactic - Test; Therapeutic
Device: best practice VTE prophylaxis — Best practice VTE prophylaxis includes sequential compression machines, compression stockings, and anticoagulants (blood thinners) when indicated.
  Arms: Prophylactic - Control

SUMMARY:
The objective of the study is to evaluate the safety and efficacy of the Adient absorbable filter for the prevention of pulmonary embolism (PE: blood clot in the lungs). PE claims the lives of over 100,000 Americans each year, more than breast cancer, traffic fatalities and HIV combined.

Pharmaceutical anticoagulation (blood thinners) that reduce blood clot formation represent the standard of care for treating patients at risk for PE. However, for people who are temporarily unable to use anticoagulants, such as those who have suffered major trauma or those who are scheduled for surgical procedures, inferior vena cava (IVC) filters are used to help protect against PE. These blood filters prevent large blood clots that originate in the deep veins of the legs (deep vein thrombosis (DVT)) from reaching your lungs causing a potentially life-threatening PE.

Conventional metal IVC filters have been proven effective at reducing the incidence of PE, however, most require retrieval. If not retrieved within a timely manner (months), they can perforate the IVC, impale nearby organs with their barbed struts, and cause blood clots.

In contrast, the Adient absorbable filter traps blood clots similar to conventional metal IVC filters, but following the 8 week protection period, the filter itself breaks down into carbon dioxide and water. Hence no filter retrieval is required and complications are less likely due to the shortened indwell time. Once blood clots are trapped in the absorbable filter, the body's thrombolytic enzymes dissolve the clots within weeks while the filter itself resorbs in 6 to 8 months. The absorbable filter is braided from absorbable suture that has been proven safe over 4 decades.

The question being addressed with the randomized controlled trial portion is whether the placement of the absorbable filter in addition to current best practice PE prevention (sequential compression machines, compression stockings, and anticoagulants when indicated) significantly reduces the incidence of clinically significant PE in high risk subjects.

The absorbable filter will be indicated for the temporary prevention of PE in patients with transient high risk for venous thromboembolism (DVT and/or PE) with or without venous thromboembolic disease and as an enhancement to pharmaceutical anticoagulation and mechanical prophylaxis.

ELIGIBILITY:
INCLUSION CRITERIA:

Aged 18 years or older

Willing to comply with the specified follow-up requirements including contrast enhanced CTs for the 9-month duration of the study

For female subjects of childbearing potential: a negative pregnancy test within 48 hours prior to the implantation procedure

For the prophylactic cohort, high risk VTE denoted by either:

Caprini score > 8 for surgical ICU, Parvizi score ≥ 150 for TKA (total knee replacement), ISS score ≥ 24 for trauma.

For the therapeutic cohort, documented VTE per the following:

Pulmonary thromboembolism when anticoagulants are contraindicated, Failure of anticoagulant therapy in thromboembolic diseases, Emergency treatment following massive pulmonary embolism where anticipated benefits of conventional therapy are reduced.

Requirement of temporary PE protection (8 weeks) based on clinical judgment

Fully informed subject or caretaker consent having executed an Institutional Review Board (IRB) or approved informed consent.

EXCLUSION CRITERIA:

Expected high VTE risk to extend beyond 8 weeks.

Vena cava filter currently implanted

History of abdominal or pelvic radiation therapy

Previous IVC filter placement/retrieval within 6 months prior to randomization

Confirmed positive blood cultures within the last 48 hours if there is bacteremia

Known sensitivity to radiographic contrast medium that cannot be adequately prophylactically pre-medicated

Known allergy or intolerance to IVC filter materials (i.e. PDSII absorbable suture)

Pregnant, lactating, or plans to become pregnant during investigation follow-up period

Renal insufficiency (GFR < 60) or requiring renal replacement therapy

IVC effective diameter (D) <16 mm or >28 mm anywhere within L1-L4, D = √(AP*Lat)

Less than 7cm from inferior-most renal vein to the iliac vein confluence

Duplication of the IVC

Any thrombus or occlusion in IVC on pre-procedural CT cavogram

Life expectancy of < 12 months

Simultaneous participation in another investigative drug or device trial that has not reached its primary endpoint

Other co-morbid condition that, in the opinion of the Investigator, could limit the subject's ability to participate in or would affect the scientific integrity of the study

Previously enrolled in a clinical investigation of the Adient filter.

For Roll In, patient has advanced heart failure or recent (6 weeks) myocardial infarction. - - -

Advanced heart failure is defined by NYHA class IV or AHA/ACC/HFSA stage D or LVEF < 40%. Subjects with MI diagnosed with ECG alone without MI history and symptoms are not excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 854 (Estimated)
Dates: Start 2023-01-27 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint - Prophylactic Cohort: incidence of new clinically significant PE | 2 weeks for asymptomatic proximal PE screening and through 8 weeks for symptomatic PE
  Clinically significant PE includes asymptomatic proximal PE screened at 2 weeks, in addition to symptomatic PE through 8 weeks post index event confirmed by computed tomography (CT) angiography. Proximal PE includes thrombus (blood clots) observed in the pulmonary trunk, main pulmonary arteries, or lobar arteries.
Primary Composite Safety Endpoint - Prophylactic Cohort: incidence of absorbable filter deployment without complications | 96 hours to 9 months depending on the safety parameter
  Potential complications include: (a) caval thrombotic occlusion within 9 months, (b) all-filter embolization within 9 months, (c) serious filter-related complications within 9 months, (d) filter placement procedural related Series Adverse Events (SAE) within the perioperative period (96 hours), (e) filter placement vascular access site SAE within the perioperative period, (f) symptomatic PE subsequent to filter deployment within 9 months.
Primary DVT Safety Endpoint - Prophylactic Cohort: incidence of all DVT post index event | 9 months overall duration
  All DVT includes both symptomatic DVT and asymptomatic DVT screened at 2 weeks, 10 weeks and 9 months.
Primary Composite Safety and Effectiveness Endpoint - Therapeutic Cohort: composite rate of technical filter placement success without complications | 9 months
  Potential complications include (a) new symptomatic PE through 8 weeks, (b) filter migration (> 2cm), (c) filter embolization, (d) caval perforation (> 5mm), (e) symptomatic caval thrombosis, and (f) any other symptomatic filter-related complication requiring invasive intervention, or filter related death.

SECONDARY OUTCOMES:
Incidence of new symptomatic PE through 8 weeks confirmed by CT angiography | 8 weeks
Miller Score for symptomatic and asymptomatic PE | 9 months
  Quantification of the occlusion of the pulmonary vascular bed from a PE.
Incidence of caval occlusion / thrombosis confirmed by CT cavogram | 10 weeks
Incidence of IVC caval stenosis and occlusion confirmed by CT cavogram | 9 months
Incidence of common femoral and iliac venous thrombosis ipsilateral to filter insertion site | 2 weeks, 10 weeks, and 9 months
  Detected on ultrasound.
Incidence of DVT | 2 weeks, 10 weeks, and 9 months
  Detected on ultrasound.
Incidence of major procedure-related or device-related adverse events | 9 months
Incidence of major bleeding | 9 months
  Major bleeding defined by International Society on Thrombosis and Haemostases.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Johnson, MD, Principal Investigator — Indiana University School of Medicine
Locations (2):
- United States (2):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - IU Health University Hospital, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elizondo G, Eggers M, Falcon M, Trevino M, Marrufo R, Perez C, Nunez E, Moreno R, Mitchell A, Sheppard A, Dria S, Jay T, Kirk R, Hovsepian D, Steele J. First-in-Human Study with Eight Patients Using an Absorbable Vena Cava Filter for the Prevention of Pulmonary Embolism. J Vasc Interv Radiol. 2020 Nov;31(11):1817-1824. doi: 10.1016/j.jvir.2020.07.021. Epub 2020 Sep 29. PMID 33008719
- [Background] Eggers M, Rousselle S, Urtz M, Albright R, Will A, Jourden B, Godshalk C, Dria S, Huang S, Steele J. Randomized Controlled Study of an Absorbable Vena Cava Filter in a Porcine Model. J Vasc Interv Radiol. 2019 Sep;30(9):1487-1494.e4. doi: 10.1016/j.jvir.2019.03.010. Epub 2019 Jun 13. PMID 31202677
- [Background] Huang SY, Eggers M, McArthur MJ, Dixon KA, McWatters A, Dria S, Hill LR, Melancon MP, Steele JR, Wallace MJ. Safety and Efficacy of an Absorbable Filter in the Inferior Vena Cava to Prevent Pulmonary Embolism in Swine. Radiology. 2017 Dec;285(3):820-829. doi: 10.1148/radiol.2017161880. Epub 2017 Jul 14. PMID 28708470
- [Background] Dria SJ, Eggers MD. In vitro evaluation of clot capture efficiency of an absorbable vena cava filter. J Vasc Surg Venous Lymphat Disord. 2016 Oct;4(4):472-8. doi: 10.1016/j.jvsv.2016.05.006. Epub 2016 Jul 25. PMID 27639002
- [Background] Eggers MD, McArthur MJ, Figueira TA, Abdelsalam ME, Dixon KP, Pageon LR, Wallace MJ, Huang SY. Pilot in vivo study of an absorbable polydioxanone vena cava filter. J Vasc Surg Venous Lymphat Disord. 2015 Oct;3(4):409-420. doi: 10.1016/j.jvsv.2015.03.004. Epub 2015 Jun 18. PMID 26992619
- [Background] Eggers MD, Reitman CA. In vitro analysis of polymer candidates for the development of absorbable vascular filters. J Vasc Interv Radiol. 2012 Aug;23(8):1023-30. doi: 10.1016/j.jvir.2012.05.039. PMID 22840802